CLINICAL TRIAL: NCT03565601
Title: Phenotypic Features and Prognostic Value of Anti-Ro52 (TRIM-21) Antibodies in Connective Tissue Diseases
Brief Title: Prognostic Value of Anti-Ro52 Antibodies in Connective Tissue Diseases (a-Ro52)
Acronym: a-Ro52
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2018/AR052-DECKER/MS
Record Dates: First submitted 2018-06-05; First posted 2018-06-21 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Connective Tissue Diseases
MeSH Terms: conditions — Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTD patients with anti-Ro52 antibodies: Connective tissue disease patients with anti-Ro52 antibodies at diagnosis
  Interventions: Other: Follow-up
- CTD patients without anti-Ro52 antibodies: Connective tissue disease patients without anti-Ro52 antibodies at diagnosis
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Clinical data, radiological data and laboratory tests follow-up

SUMMARY:
Anti-Ro52 autoantibodies can be detected in patients with several autoimmune diseases. Clinical significance of anti-Ro52 is controversial. The presence of anti-Ro52 may be a factor associated with disease severity (interstitial lung disease, vasculopathy) and cancers. The aim of this study is to assess interstitial lung disease and vasculopathy prevalence and severity, cancers occurence and others clinical features of connective tissue disease patients with anti-Ro52 autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* Connective tissue disease (differenciated or not)
* Presence of anti-Ro52 antibodies at diagnosis

Exclusion Criteria:

* Healthy subjects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with connective tissue disease (differenciated or not) and anti-Ro52 antibodies (as single specificity or associated with other autoantibody specificities) at diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
ILD prevalence | baseline (J0)
  Clinical (cough, dyspnea) and/or radiological (tomodensitometry) data

SECONDARY OUTCOMES:
ILD severity | baseline (J0)
  PFT (pulmonary function test): FVC, FEV1, DLCO (percentages of predicted values)
Vasculopathy occurence | baseline (J0) and follow-up
  Raynaud disease, digital ulcers or gangrene
Cancer occurence | baseline (J0) and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Roland JAUSSAUD, Pr, Principal Investigator — Central Hospital, Nancy, France; Paul DECKER, MR, Study Director — Central Hospital, Nancy, France
Locations (4):
- France (4):
  - Central Hospital, Dijon
  - Central Hospital, Lille
  - Private Hospital, Metz
  - Central Hospital, Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghillani P, Andre C, Toly C, Rouquette AM, Bengoufa D, Nicaise P, Goulvestre C, Gleizes A, Dragon-Durey MA, Alyanakian MA, Chretien P, Chollet-Martin S, Musset L, Weill B, Johanet C. Clinical significance of anti-Ro52 (TRIM21) antibodies non-associated with anti-SSA 60kDa antibodies: results of a multicentric study. Autoimmun Rev. 2011 Jul;10(9):509-13. doi: 10.1016/j.autrev.2011.03.004. Epub 2011 Apr 5. PMID 21447407
- [Background] Lee AYS. A review of the role and clinical utility of anti-Ro52/TRIM21 in systemic autoimmunity. Rheumatol Int. 2017 Aug;37(8):1323-1333. doi: 10.1007/s00296-017-3718-1. Epub 2017 Apr 17. PMID 28417151
- [Background] Hudson M, Pope J, Mahler M, Tatibouet S, Steele R, Baron M; Canadian Scleroderma Research Group (CSRG); Fritzler MJ. Clinical significance of antibodies to Ro52/TRIM21 in systemic sclerosis. Arthritis Res Ther. 2012 Mar 6;14(2):R50. doi: 10.1186/ar3763. PMID 22394602
- [Background] Gunnarsson R, El-Hage F, Aalokken TM, Reiseter S, Lund MB, Garen T; Norwegian MCTD study group; Molberg O. Associations between anti-Ro52 antibodies and lung fibrosis in mixed connective tissue disease. Rheumatology (Oxford). 2016 Jan;55(1):103-8. doi: 10.1093/rheumatology/kev300. Epub 2015 Aug 28. PMID 26320136
- [Background] Murng SHK, Thomas M. Clinical associations of the positive anti Ro52 without Ro60 autoantibodies: undifferentiated connective tissue diseases. J Clin Pathol. 2018 Jan;71(1):12-19. doi: 10.1136/jclinpath-2015-203587. Epub 2017 Jun 29. PMID 28663326
- [Background] Reiseter S, Gunnarsson R, Mogens Aalokken T, Lund MB, Mynarek G, Corander J, Haydon J, Molberg O. Progression and mortality of interstitial lung disease in mixed connective tissue disease: a long-term observational nationwide cohort study. Rheumatology (Oxford). 2018 Feb 1;57(2):255-262. doi: 10.1093/rheumatology/kex077. PMID 28379478
- [Background] Bauhammer J, Blank N, Max R, Lorenz HM, Wagner U, Krause D, Fiehn C. Rituximab in the Treatment of Jo1 Antibody-associated Antisynthetase Syndrome: Anti-Ro52 Positivity as a Marker for Severity and Treatment Response. J Rheumatol. 2016 Aug;43(8):1566-74. doi: 10.3899/jrheum.150844. Epub 2016 Jun 1. PMID 27252419